CLINICAL TRIAL: NCT02784626
Title: The Influence of Intraoperative Sedative on Postoperative Pain in Total Knee Arthroplasty Under Spinal Anesthesia: Comparison Between Dexmedetomidine and Propofol
Brief Title: Intraoperative Sedatives and Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B-1603/339-005
Record Dates: First submitted 2016-05-22; First posted 2016-05-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Arthritis, Degenerative
Keywords: Dexmedetomidine; Propofol; Pain, Postoperative
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients who received dexmedetomidine during the operation
  Interventions: Drug: Dexmedetomidine
- Propofol (Experimental): Patients who received propofol during the operation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Intraoperative sedation using dexmedetomidine
  Arms: Dexmedetomidine
Drug: Propofol — Intraoperative sedation using propofol
  Arms: Propofol

SUMMARY:
In this study, based on the hypothesis that dexmedetomidine administered intraoperatively for sedation can reduce postoperative pain than that of propofol, the investigators examined the ability of dexmedetomidine to reduce postoperative pain in in patients undergoing the total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty
* Age: 20 - 80 yrs

Exclusion Criteria:

* ASA classification ≥ 3
* Patient who do not want sedation during the surgery
* Patient who wants general anesthesia
* Cardiovascular disease
* Liver dysfunction
* Renal dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Postoperative 24 hours
  Postoperative pain score at postoperative 24 hours

SECONDARY OUTCOMES:
Rescue analgesics | Postoperative 24 hours
  Amount of rescue analgesics administered during 24 hours postoperatively
Rescue analgesics | Postoperative 48 hours
  Amount of rescue analgesics administered during 48 hours postoperatively
Visual analogue scale | Postoperative 48 hours
  Postoperative pain score at postoperative 48 hours

OTHER OUTCOMES:
Nausea and vomiting | Postoperative 24 hours
  Incidence of nausea and vomiting during 24 hours postoperatively
Nausea and vomiting | Postoperative 48 hours
  Incidence of nausea and vomiting during 48 hours postoperatively
Antiemetics | Postoperative 24 hours
  Amount of antiemetics administered during 24 hours postoperatively
Antiemetics | Postoperative 48 hours
  Amount of antiemetics administered during 48 hours postoperatively
Patient's satisfaction | Postoperative 48 hours
  Patient's satisfaction with the pain management using a visual analogue scale (0 = very unsatisfied, 10 = completely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No